CLINICAL TRIAL: NCT03517579
Title: Personalized Treatment Planning for Radio-iodine Therapy of Thyroid Disease
Brief Title: Personalized Treatment in Thyroid Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00157150
Record Dates: First submitted 2018-04-03; First posted 2018-05-07 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Thyroid Cancer; Graves Disease
MeSH Terms: conditions — Thyroid Neoplasms; Graves Disease

STUDY DESIGN:
Intervention Model Description: This is a pilot experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Project (Experimental): It is a Pilot study of 10 persons
  Interventions: Device: Cervical Collar Therapy Indicator (COTI)

INTERVENTIONS:
Device: Cervical Collar Therapy Indicator (COTI) — Study Device; The CoTI has 3 components;
  * A collar unit: a gamma detector wrapped around a body part-neck in this case and contains a scintillating crystal and a silicon photomultiplier. The photon pulse signal is then converted to digital signals (measuring the counts per second). Usually two detectors are placed in specified positions.
  * A cable that connects the collar unit to the Control Unit
  * A control unit that collects the signals and transmits it wirelessly to a hand-held computer tablet.
  Two types of collar devices will be used: the lower activity and the medium activity
  1. Lower activity collar for patients with Graves' disease as well as diagnostic I-123 scan in thyroid cancer patients. These patients typically receive 0.2-1.2 m Ci of I-123/I-131.
  2. Medium activity collar for Patients with thyroid cancer after 131-I ablation, for which patients typically receive 30-100 mci of I-131.

SUMMARY:
The Collar Therapy Indicator (CoTI) (A device that is placed in collar around the neck resembling a turtle neck sweater collar with a wire and recording box) has been shown in a single small previously published experience to provide data regarding radioiodine exposure that correlates with conventional methods of measuring I-123 and I-131 uptakes after diagnostic dose administration and/or therapy for thyroid disorders. We hypothesize that the device's continuous measurement capability will permit more accurate estimates of radiation exposure to thyroid tissue than conventionally employed methods assessing fractional uptake at one or a few time points. It may also provide information about the extent of variability in the absorbed radiation dose among patients with thyroid cancer and hyperthyroidism. By providing more complete information about individual patient's exposures, it will facilitate more accurate estimation of the administered I-131 dose requirements for control of hyperthyroidism and thyroid remnant ablation while reducing the need for repeated visits to the clinic for dosimetry measurements. The aims of our project include the following: (1)To compare quantitative imaging-derived thyroid time activity curve to that obtained using the CoTI and to determine the extent to which there is variability in radiation dose predicted using conventional methods to that predicted from measurement of the full Time-Activity Curve (TAC).(2) Evaluate the uptake and clearance kinetics across the 5 patients in each category as proof of principle for a potential larger trial to investigate use of this device in optimizing the administered doses of radioactive iodine to achieve therapeutic goals while minimizing risks of comorbidities, such a post-radioiodine hypothyroidism in patients with Graves' disease.(3)Evaluate patient experience, convenience, and discomfort in using the CoTI device with a survey instrument.

DETAILED DESCRIPTION:
Radioiodine treatment for thyroid disorders represented an early example of individualized medicine. Since its introduction 80 years ago, the therapeutic I-131 dosage has usually been tailored to individual patient requirements based on the uptake of a tracer radioiodine dose. Various techniques have been employed to estimate the administered dose of I-131 for optimal therapeutic benefit. Estimated exposure has typically been extrapolated from the results of activity measurements at one or two time points, e.g., at 4 and 24 hours. We now know that treatment of hyperthyroid Graves' disease with these methods lead to a 13-25% rate of failure to cure hyperthyroidism and a 46-80% rate of long-term hypothyroidism in cured patients. Similarly, such relatively crude dosimetry doubtless result in significant overtreatment in the case of remnant ablation for differentiated thyroid cancer.

For patients with differentiated thyroid cancer requiring remnant ablation, the administered activity has, in most cases, been derived empirically, ranging between 30-100 mci. The high success rates in ablating remnant thyroid tissue implies that many patients are still treated with higher 131-I doses than required, with potential side effects, such as radiation sialadenitis.

Pilot Study Rationale; Our overall objective is to provide the optimal dose to each patient. This study will apply a novel "wearable" radiation detection technology to determine continuous cervical measurements over days following tracer radioiodine administration will provide information that permits the tailoring of subsequent therapeutic radioiodine doses more precisely to improve clinical outcomes, as described above.

The actual therapeutic dose decisions in this pilot trial, however, will not be based on the collar device measurements. Patients with Graves' disease will receive 180-200 µCi I-131 per gram of estimated gland mass based on the conventional method of dose calculation, based on a 24-hour % uptake and gland volume. Most patients with thyroid cancer would receive the 30 mCi dose for remnant ablation prior to the placement of the COTI device, as per the American Thyroid Association (ATA) guidelines.

STUDY DESIGN AND METHODS This will be an unmasked prospective pilot study involving patients with Graves' disease (Group I) and differentiated thyroid cancer (Group II). Five patients in each group will have radiation activity measurements using the COTI devise. All persons in the study will receive 131-I treatment based on the current standards of care for dose estimation.

Study Device; The CoTI has 3 components;

* A collar unit: a gamma detector wrapped around a body part-neck in this case and contains a scintillating crystal and a silicon photomultiplier. The photon pulse signal is then converted to digital signals (measuring the counts per second). Usually two detectors are placed in specified positions.
* A cable that connects the collar unit to the Control Unit
* A control unit that collects the signals and transmits it wirelessly to a hand-held computer tablet.

Two types of collar devices will be used: the lower activity and the medium activity

1. Lower activity collar for patients with Graves' disease as well as diagnostic I-123 scan in thyroid cancer patients. These patients typically receive 0.2-1.2 m Ci of I-123/I-131.
2. Medium activity collar for Patients with thyroid cancer after 131-I ablation, for which patients typically receive 30-100 mci of I-131.

Study Population;

* Group I: Patients with diffuse toxic goiter (Graves' disease) diagnosed clinically with no prior history of radioiodine treatment.
* Group II: Patients with differentiated epithelial thyroid cancer who are s/p total thyroidectomy and candidates for remnant ablation based on ATA guidelines.

IRB approval and HIPPA regulations; Since it is a project involving a medical device which will be applied to the patients' neck, it will require the following;

1. Institutional Review Board (IRB) regular approval.
2. Registry into ClinicalTrials.gov.
3. Appropriate forms and consent process for the patients. The recruitment of subjects for the study;

   * Informed consent including the benefits and the risks of the Collar device (CoTI) will be obtained.
   * Confidentiality agreement would be signed regarding the CoTI and its application.
   * Demographic, clinical and tumor characteristics of the participants will be obtained, as outlined below.
   * The instructions on the application CoTI will be provided in detail.
   * Instructions regarding communication in the event of any difficulties will be provided.

Preparation the patient;

1. The patients will be prepared by general standards of care prior to CoTI placement. For patients with Graves' disease, any thionamide anti-thyroid meds will be stopped 3-5 days prior to I-123 diagnostic dose administration. After obtaining written consent, a venous blood sample will be obtained for work for requisite laboratory evaluation for baseline labs, as outlined below, and in women, for a pregnancy test. A (low activity) CoTI device will be placed under supervision and then adjusted for comfort and optimal activity measurement as a trial and then removed. Background activity of the patient, a phantom, and the device itself will be measured. After administration of I-123, an initial uptake at time 0 will be obtained. The CoTI device will then be placed and the patient will be asked to return to the clinic at scheduled imaging times for Group I. Anatomical localization of the CoTI in all patients will be standardized by pen markings.
2. Patients with Graves' disease, who will be administered 200 µCi of I-131 and fitted with a low-activity CoTI device after administration of the dose. Background activity of the patient, a phantom and the device itself will be measured prior to placement of the device. After administration of I-131, an initial uptake at time 0 will be obtained. The CoTI device will then be placed and the patient will be asked to come back at scheduled imaging times for Group II. Anatomical localization for the CoTI for all patients will be standardized by markings.
3. Patients with differentiated thyroid cancer will be placed on a low iodine diet for one week. Recombinant TSH will be administered on days 1 and 2 (typically Monday and Tuesday), and the diagnostic I-123 dosage will be administered on day 2. As per the protocol standard of care, the diagnostic whole-body scan is done on day 3 and the I-131 dose for I-131 ablation (30-100 mci) is administered on day 4.

After obtaining written consent, venous blood sample will be obtained for work for requisite laboratory evaluation for baseline labs as outlined below, including in women, a pregnancy test prior to the I-131 remnant ablation dose. The (medium activity) CoTI device will be placed under supervision and then adjusted for convenience as outlined above. Background activity of the patient, a phantom, and the device itself will be measured. After administration of I-131, an initial uptake at time 0 will be obtained. The CoTI device will then be placed and the patient will be asked to come back at scheduled imaging times for Group II. Anatomical localization for the CoTI for all patients will be standardized by markings.

Scheduled Imaging times; Group I - Persons with Graves' Disease

1. After I-123 diagnostic dose - A planar image with a pinhole collimator at time 06.00 hours.

   - An uptake only measurement at time 12.00 hours using the uptake probe.
   * An uptake only measurement (with the probe) at time 24.00 hours.
   * The counts from the handheld device connected to the CoTI would be obtained at similar times as above with one additional time point of 18.00 hours i.e. 0, 6, 12, 18 and 24 hours.
2. After administration of 200 µCi of I-131 dose

   - A first SPECT image would be performed at 6 hours after I-131 dose.
   * A Second SPECT image (with a low dose CT for quantification and attenuation correction) would be performed at 24 hours after I-131 dose.
   * A third SPECT image at 48 hours.
   * A fourth SPECT image at 72 hours.
   * The counts from the handheld device connected to the CoTI would be obtained at similar times as above with one additional time point of 96.00 hours i.e. 6, 24, 48, 72 and 96.

   Group II - Persons with Thyroid Cancer

   -A SPECT image would be performed at 24 hours (with low dose CT for quantification and attenuation correction) after I-131 therapy.

   -A second SPECT image at 48 hours.

   -A third SPECT image at 72 hours (with low dose CT for quantification and attenuation correction).

   A final SPECT CT image (with low dose CT for quantification and attenuation correction) at day 7 post therapy.

   - The counts from the handheld device connected to the CoTI would be obtained at similar times as above with one additional time point of 96.00 hours i.e. 24, 48, 96 and day 7.

   Data collection, periodic follow up; • Baseline data will include age, gender, BMI; duration of autoimmune thyroid disease and/or differentiated thyroid cancer, History/details of thyroid cancer (stage, Fine Needle Aspiration (FNA) findings, final tumor histopathology, presence of lymph node metastasis thyroglobulin levels- baseline and stimulated, preoperative ultrasound findings, extent of surgery); presence of co-morbidities, details of autoimmune thyroid disease (prior anti-thyroid regimen including duration of discontinuation, thyroid function tests (free thyroxine, free triiodothyronine, TSH), thyroid antibodies, and thyroid stimulating immunoglobulins ), duration and history of levothyroxine therapy (in cases with thyroid cancer), results of neck and thyroid ultrasound, measured neck circumference prior to application of device, quality of life scores as measured by a questionnaire. Imaging data would be acquired as outlined above Statistical Analysis; Descriptive data will be outlined for all the participants tabulating the variables as determined. The intrapatient variability as well as accuracy and precision of the device will be obtained individually for Group I and Group II patients. The correlation (non-parametric) Spearman correlation coefficient will be obtained to assess the relationship between the uptake and findings as obtained by the collar device and conventional methods of uptake measurement.

ELIGIBILITY:
Inclusion Criteria:

* Group I

  * Patients with Graves' disease confirmed by laboratory testing.
  * Patients able to understand English and able to follow instructions. Group II
  * Patients with intermediate and high risk differentiated thyroid cancer requiring radioiodine remnant ablation or moderately high dose I-131 for treatment of residual cervical disease.
  * Persons able to understand simple English and able to follow instructions.

Exclusion Criteria:

* Patients with diseases involving cervical spine, such as spondylosis and severe degenerative joint disease.
* Pregnant Women, elderly and persons unable to understand simple instructions

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-12-11 (Actual); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the Variability in radioiodine kinetics for patients with thyroid cancer and graves disease | 6-9 months
  Radioactive iodine uptake at different time points will be taken over a 24 hour period (7 days for thyroid cancer) and then the Area Under the Curve (AUC) will be Plotted.The AUC would then be correlated with the 24 hour uptake in Graves and day 7 uptake for thyroid cancer.We will use non-parametric tests to measure the correlation

SECONDARY OUTCOMES:
Validation of the device as an enhancement of quantitative measurements in patients with Graves disease and thyroid cancer | 9-12 months
  Using SPECT-CT (the best current method for quantitative measurements of the thyroid uptake) ,we will compute the uptake of I-131 at different time points (as mentioned in the protocol) and correlate it with the AUC (computed by the COTI device) and see the degree of congruity. In the case of graves disease patients, the 6 hour and 24 hour uptake (standard of care) would be measured against the COTI AUC

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Santhanam, MBBS, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Other than the study researchers, the data will not be shared with anyone else

REFERENCES:
- [Background] Ladenson PW. Precision Medicine Comes to Thyroidology. J Clin Endocrinol Metab. 2016 Mar;101(3):799-803. doi: 10.1210/jc.2015-3695. Epub 2016 Feb 23. PMID 26908108
- [Result] Brinks P, Van Gils K, Kranenborg E, Lavalaye J, Dieckens D, Habraken JBA. Measuring the actual I-131 thyroid uptake curve with a collar detector system: a feasibility study. Eur J Nucl Med Mol Imaging. 2017 Jun;44(6):935-940. doi: 10.1007/s00259-016-3595-y. Epub 2016 Dec 17. PMID 27988801
- [Derived] Santhanam P, Solnes L, Nath T, Roussin JP, Gray D, Frey E, Sgouros G, Ladenson PW. Real-time quantitation of thyroidal radioiodine uptake in thyroid disease with monitoring by a collar detection device. Sci Rep. 2021 Sep 16;11(1):18479. doi: 10.1038/s41598-021-97408-y. PMID 34531443